CLINICAL TRIAL: NCT01574742
Title: A Single Center, Open Label Study Assessing the Feasibility, Safety and Therapeutic Effect of Minocycline in Adult Patients With Diagnosis of Unipolar Depression.
Brief Title: Open Study Assessing the Feasibility of Minocycline in Patients With Unipolar Depression
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0007-12-SHA
Record Dates: First submitted 2012-04-09; First posted 2012-04-10 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-04

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minocycline (Experimental): Minocycline 200 mg/day (2X100 mg) from day 1 to day 3 and Minocycline 400 mg/day (2X200mg) form day 4 until termination visit (day 35)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 200 mg/day (2X100 mg) from day 1 to day 3 and Minocycline 400 mg/day (2X200mg) form day 4 until termination visit (day 35)
  Other Names: Minoclin

SUMMARY:
A single center, open label study assessing the feasibility, safety and therapeutic effect of Minocycline in adult patients with diagnosis of unipolar depression. Up to 30 patients diagnosed with unipolar depression that are in a current depressive episode. The patients will be of all racial, ethnic and gender categories, ranging from 18 to 68 years of age, and have HDRS-21≥20. All subjects will continue to take their treatment with antidepressant medications for the duration of the study. All subjects are prescribed minocycline 200 mg/day orally (2X100 mg) for the first 3 days. than, all subjects are prescribed minocycline 400 mg/day orally (2X200 mg) from day 4 until termination visit (day 35). The primary objective of this study is to assess the therapeutic effect of Minocycline in unipolar depression.

The secondary objectives of this study are to assess the therapeutic effect, the feasibility and safety of Minocycline in unipolar depression.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients and inpatients
2. Men and women 18-68 years of age.
3. Primary DSM-IV diagnosis of Depression, single or recurrent episode confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV), with the additional requirements of a current episode ≥4 weeks and CGI-S ≥4.
4. Total HDRS-21 ≥20 and Item 1 score ≥2 at the screening visit.
5. The patient did not respond to at least one antidepressant medication given for an accepted dose and duration.
6. Capable and willing to provide informed consent
7. Able to adhere to the treatment schedule.

   -

Exclusion Criteria:

1. Depression secondary to a general medical condition.
2. History of substance abuse or dependence within the past 6 month (except opioids, nicotine and caffeine).
3. All antidepressant medications, must have been in stable dosage for at least 3 weeks prior to entry into the study, with no anticipation of change over the duration of the study.
4. Use of any medication(s) listed on the Excluded medication list within the time that mansion for each medication on the list.
5. Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features • Bipolar disorder • Eating disorder
6. Subjects who were taking a known contraindication to minocycline treatment.
7. Subjects who had received treatment with minocycline or β-lactam antibiotics in the preceding half year before study entry.
8. Present suicidal risk as assessed by the investigator or significant suicide risk based on HDRS-21 item 3 score of 3 or 4 or a history of attempted suicide in the last 6 month
9. Known or suspected pregnancy or women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.(if using oral contraceptives, during the minocycline treatment, subject should use an additional contraceptives), or women who are breastfeeding
10. Patients with severe hepatic or renal insufficiency.

    -

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | from baseline (day 1) to termination (day 35)
  The change in Scale for Depression (HDRS-21) score from baseline to the end of the study (visit 4 - day 35) where response is defined as ≤50% reduction in HDRS-21 score from baseline.

SECONDARY OUTCOMES:
Depression symptoms - CGI | from baseline (day 1) untill termination visit (day 35)
  The change in Clinical Global Impression Scale (CGI) from baseline to the end of the study.
depression symptoms - (QIDS-SR) | from baseline (day 1) untill termination visit (day 35)
  The change in Quick Inventory of Depressive Symptology -self report (QIDS-SR) from baseline to the end of the study.
depression symptoms - HDRS-21 | from baseline (day 1) untill termination visit (day 35)
  Remission rates after 5 weeks of Minocycline treatment, where remission is defined as HDRS-21 score <10.
Safety | frpm baseline (day 1) untill the termination visit (day 35)
  Safety Evaluation: Tolerability of Minocycline as defined by maintained subject baseline, pre-treatment, physical and neurological examinations and lack of significant increase in suicide ideation measured by:
  * Vital signs
  * Physical and neurological examination
  * Any other adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, PhD, Principal Investigator — Shalvata Medical Health Center
Locations (1):
- Shalvata Medical Health Center, Hod HaSharon, Israel